CLINICAL TRIAL: NCT02902432
Title: A Trial of Endostar in Patients With Carcinoma of the Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China International Medical Foundation (Other)
Collaborators: Chinese Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Ping Liu, Attending doctor in oncology, China International Medical Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChinaIMF
Record Dates: First submitted 2016-08-12; First posted 2016-09-15 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: endostar; cisplatin
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — endostar protein; Endostatins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCCHN (Placebo Comparator): patients with advanced squamous cell carcinoma of the head and neck.IMRT.
  Interventions: Drug: Endostar
- SCCHN-Endostar (Experimental): patients with advanced squamous cell carcinoma of the head and neck.Endostar will be continuously intravenous pumped (7.5 mg/m2) for 14 days (d1-d14) during chemotherapy and for 5 days/week(d-5-d-1, d3-d7, d10-d14, d17-d21)during IMRT.
  Interventions: Drug: Endostar

INTERVENTIONS:
Drug: Endostar — The patients will be randomized to CRT arm and CRT+Endostar arm. All patients will receive one cycles of induction chemotherapy, intensity modulated radiation therapy (IMRT) with weekly cisplatin and 3 cycles of chemotherapy after IMRT.
  Other Names: recombinant human endostatin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant human endostatin（continuously-pumped）combined with chemoradiotherapy in patients with advanced squamous cell carcinoma of the head and neck. The patients will be randomized to concurrent radiotherapy (CRT) arm and CRT + Endostar arm. All patients will receive one cycles of induction chemotherapy, intensity modulated radiation therapy (IMRT) with weekly cisplatin and 3 cycles of chemotherapy after IMRT. Treatment cycles will be repeated every 21 days for a maximum of 4 cycles. In CRT + Endostar arm, Endostar will be continuously intravenous pumped (7.5 mg/m2) for 14 days (d1-d14) during chemotherapy and for 5 days/week (d-5-d-1, d3-d7, d10-d14, d17-d21) during IMRT.

DETAILED DESCRIPTION:
The patients will be randomized to CRT arm and CRT + Endostar arm. All patients will receive one cycles of induction chemotherapy, intensity modulated radiation therapy (IMRT) with weekly cisplatin and 3 cycles of chemotherapy after IMRT. Treatment cycles will be repeated every 21 days for a maximum of 4 cycles. In CRT + Endostar arm, Endostar will be continuously intravenous pumped (7.5 mg/m2) for 14 days (d1-d14) during chemotherapy and for 5 days/week (d-5-d-1, d3-d7, d10-d14, d17-d21) during IMRT.

Prior to enrollment in this study and while the patient is receiving the therapy, routine tests, ECG, head and neck CT scan and MRI will be performed to check the body's response to the treatment. Further more, before and after the treatment, the circulating endothelial cells (CECs), endothelial progenitor cells (CEPs), vascular endothelial growth factor (VEGF), Cancer embryo antigen (CEA), Neuron-specific enolase (NSE) in blood and Microvessel density (MVD), hypoxia-inducible factor-1a (HIF-1a), P53, VEGF, Survivin in pathological specimens will be tested.

Patients with progressive disease or intolerable side effects will be removed from the study. Patients with stable disease or tumor response will continue therapy for a maximum of 4 cycles.

Primary outcome: The response rate (RR), the clinical benefit rate (CBR), time of tumor progression (TTP).

Secondary outcomes: The quality of life (QOL)，Safety and Tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unrespectable or postoperative recurrent squamous cell carcinoma of the head and neck;
* No prior radiation or chemotherapy and biotherapy before;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.Life expectancy greater than 3 months;
* Patients must have adequate bone marrow function:

  * Platelets ≥ 80×109/L
  * Hemoglobin ≥100 g/L
  * Absolute NeutrophilCount ≥1.5×109/L
  * white blood cell≥ 3.5×109/L
* Patients must have adequate liver and renal function:

  * Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) < 2.5 × upper limit of normal
  * Alkaline phosphatase < 2.5 × upper limit of normal
  * Total bilirubin < 1.5 mg/dL
  * Creatinine <1.5 mg/dL× upper limit of normal
* A cardiac ejection fraction > 50%;
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Participation in any investigational drug study within 4 weeks preceding the start of study treatment;
* Age ≤18 or ≥75 years of Age;
* Pregnant or breastfeeding women;
* Serious, uncontrolled, concurrent infection(s) requiring antibiotics;
* Clinically apparent central nervous system metastases or carcinomatous meningitis;
* Treatment for other carcinomas within the last 3 months;
* Patient unable or not willing to perform all study related biopsies and blood draws for exploratory endpoints will not be enrolled on study as all study related procedures are mandatory;
* Patients with clinically significant cardiac disease (New York Heart Association Classification III or IV and cardiac arrhythmias not well controlled with medication), or myocardial infarction within the previous six months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12-20 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (Mon); PFS, According to RECIST v1.1 | up to 40 months
  Time of tumor progression in patients with head and neck squamous cell carcinoma

SECONDARY OUTCOMES:
Quality of life (QOL); Scores range from 0 to 5 | up to 40 months
  Quality of life (QOL) in cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: ping liu, doctor, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- the Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided